CLINICAL TRIAL: NCT01359813
Title: Effects of Albumin Administration in Septic Cirrhotic Patients With Child > 8 Unrelated to Spontaneous Bacterial Peritonitis on Renal Function and Survival: A Multicenter Randomized Controlled Trial Comparing Use and Non-use of Human Albumin (Vialebex ®)
Brief Title: Albumin Administration in Cirrhotic Patients With Bacterial Infection and a Systemic Inflammatory Response Syndrome Unrelated to Spontaneous Bacterial Peritonitis
Acronym: ALB-CIRINF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: decision of independent monitoring committee:Risk of death at 3 months higher in Albumin group than in control group, without reaching significance level.
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N/2008/51
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2010-07

CONDITIONS: Cirrhosis; Sepsis; Renal Failure
MeSH Terms: conditions — Fibrosis; Sepsis; Renal Insufficiency | interventions — Serum Albumin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual treatment (No Intervention): intravenous injection of Human Albumin. 1,5g/kg on first day and 1g/kg on third day
- Human Albumin (Experimental): 1,5g/kg on first day and 1g/kg on third day.
  Interventions: Drug: Human Albumin

INTERVENTIONS:
Drug: Human Albumin — Administration: 1,5 g/kg at Day 1 and 1g/kg at Day 3 In case of a new infection appears in the 3 months, the same doses will be administrated.
  Arms: Human Albumin

SUMMARY:
Patients with cirrhosis present an increased susceptibility to bacterial infections. Spontaneous bacterial peritonitis (SBP) is the most frequent infection and induces severe circulatory dysfunction associated with renal failure in about 30% of cases. Renal failure is a reliable surrogate marker of in-hospital mortality in patients with SBP or with non-SBP infections. Albumin, as an adjuvant to antibiotherapy reduces significantly the rate of renal failure, in-hospital mortality, and overall mortality (Sort P, et al. NEJM 1999). However, little is known regarding the effect of albumin administration in patients with non-SBP infections. Two recent prospective studies demonstrated that non-SBP infections are associated with impairment of the effective circulating volume and precipitate renal failure whatever the presence of ascites.

The aim of this randomized clinical trial is to evaluate the effects of albumin, associated with appropriate antibiotic therapy, on occurrence or deterioration of renal failure and survival in septic (SIRS criteria required) cirrhotic patients with non-SBP infections and presenting with a Child-Pugh score > 8.

DETAILED DESCRIPTION:
* Cirrhosis defined by clinical, laboratory or ultrasonographic findings
* Child-Pugh > 8
* Sepsis defined by the presence of proved or suspected infection with two of the four SIRS (systemic inflammatory response syndrome) criteria (Wong F, et al. Sepsis in cirrhosis: report on the 7th meeting of the international ascites club. Gut 2005)
* Creatinine < 160 µmol/L

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis defined by clinical, laboratory or ultrasonographic findings
* Child-Pugh > 8
* Sepsis defined by the presence of proved or suspected infection with two of the four SIRS (systemic inflammatory response syndrome) criteria (Wong F, et al. Sepsis in cirrhosis: report on the 7th meeting of the international ascites club. Gut 2005)
* Creatinine < 160 µmol/L
* Written informed consent
* Absence of the exclusion criteria

Exclusion Criteria:

* Spontaneous bacterial peritonitis
* Difficult to treat infections such as : endocarditis, septic arthritis, osteomyelitis
* Heart insufficiency (YHA III-IV)
* Digestive bleeding during the week preceding the study
* Septic shock
* Hepatocellular carcinoma : stage D
* Use of antibiotics during the week preceding the study, except noroxin used for long-term antibioprophylaxy
* Diseases which can influence the short term survival

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2008-12; Primary Completion 2011-09 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Renal failure rate | at 3 months
  Occurrence or deterioration of renal failure at 3 months

SECONDARY OUTCOMES:
In-hospital and at 3-month mortality | during hospitalization and 3-month mortality

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Thevenot, PH, Principal Investigator — CHU de Besançon
Locations (35):
- France (35):
  - CHU, Amiens
  - CHU, Angers
  - CHBM, Belfort
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Hôpital Jean Verdier, Bondy
  - CHU, Bordeaux
  - CHU, Brest
  - CHU, Caen
  - Hôpital Antoine Béclère, Clamart
  - Centre Hospitalier universitaire, Clermont-Ferrand
  - Hôpital Beaujon, Clichy
  - CHIC, Créteil
  - CHU, Dijon
  - Centre Hospitalier, Dunkirk
  - CH Francilien, Évry
  - CH, Gonesse
  - CHU, Grenoble
  - CH, Lens
  - CHU, Lille
  - Centre Hospitalier Universitaire, Marseille
  - Centre Hospitalier, Maubeuge
  - Centre Hospitalier Universitaire, Nancy
  - CHU, Nice
  - CHR, Orléans
  - CHU Tenon, Paris
  - Hôpital Henri Mondor, Paris
  - Hôpital Saint Antoine, Paris
  - CHU, Pau
  - CHU, Reims
  - CHU, Rouen
  - CH, Saint-Brieuc
  - CHU, Toulouse
  - CH, Tourcoing
  - Centre Hospitalier régional Universitaire, Tours
  - Centre Hospitalier, Vesoul

REFERENCES:
- [Derived] Thevenot T, Bureau C, Oberti F, Anty R, Louvet A, Plessier A, Rudler M, Heurgue-Berlot A, Rosa I, Talbodec N, Dao T, Ozenne V, Carbonell N, Causse X, Goria O, Minello A, De Ledinghen V, Amathieu R, Barraud H, Nguyen-Khac E, Becker C, Paupard T, Botta-Fridlung D, Abdelli N, Guillemot F, Monnet E, Di Martino V. Effect of albumin in cirrhotic patients with infection other than spontaneous bacterial peritonitis. A randomized trial. J Hepatol. 2015 Apr;62(4):822-30. doi: 10.1016/j.jhep.2014.11.017. Epub 2014 Nov 21. PMID 25463545